CLINICAL TRIAL: NCT00285233
Title: An Open-label Pilot Study of Delayed Mycophenolate Mofetil Instead of Tacrolimus Combined With Anti-thymocyte Globulin, Daclizumab, Etanercept, and Sirolimus in Single-donor, Solitary Islet Allograft Recipients With Type 1 Diabetes
Brief Title: Delayed Mycophenolate Mofetil in Single-Donor Islet Allotransplantation in Type 1 Diabetes
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Roche Pharma AG (Industry); Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0006M55241
Record Dates: First submitted 2006-01-30; First posted 2006-02-01 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-07

CONDITIONS: Type 1 Diabetes; Hypoglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Biological: Allogeneic islets of Langerhans transplant

INTERVENTIONS:
Biological: Allogeneic islets of Langerhans transplant — Allogeneic islets of Langerhans transplant
  Other Names: Islet transplant

SUMMARY:
The objective of this study is to assess the safety and efficacy of islet allotransplantation for the reestablishment of stable glycemic control in patients with type 1 diabetes, using anti-thymocyte globulin induction immunosuppression with sirolimus, mycophenolate mofetil and low dose tacrolimus maintenance immunosuppression.

DETAILED DESCRIPTION:
To assess the safety and efficacy of a new single-donor islet allotransplant protocol focusing on minimization of ischemic damage by the two-layer pancreas preservation technique, attenuation of posttransplant nonspecific inflammatory responses by etanercept and anti-thymocyte globulin, deletion/inactivation of autoreactive T cells by anti-thymocyte globulin and daclizumab induction immunotherapy, and potent yet non-diabetogenic maintenance immunosuppression with sirolimus and delayed mycophenolate mofetil instead of tacrolimus for the reestablishment of stable glycemic control in recipients with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Primary islet allotransplant
2. Type 1 diabetes mellitus, complicated by at least one of the following situations that persist despite intensive efforts in close cooperation with their diabetes care team:

   1. Metabolic lability/instability;
   2. Reduced awareness of hypoglycemia;
   3. Persistently poor glucose control (as defined by HgbA1c>10% at the end of six months of intensive management efforts with the diabetes care team);
   4. Progressive secondary complications.
3. Age 18 and older
4. Able to give written informed consent

Exclusion Criteria:

1. Known hypersensitivity to rabbit proteins.
2. Presence of history of panel-reactive anti-HLA antibodies (>10%).
3. Insufficient cardiovascular reserve.
4. Creatinine clearance <60 mL/min/m2.
5. Portal hypertension, abnormal liver enzyme tests, or history of significant liver disease.
6. History of malignancy within 5 years.
7. Active peptic ulcer disease.
8. Severe unremitting diarrhea or other gastrointestinal disorders potentially interfering with the ability to absorb oral medications.
9. Pregnancy or breast-feeding.
10. Active infections.
11. Serological evidence of infection with HIV, or HBsAg or HCVAb positive within the previous 12 months prior to transplantation.
12. Negative screen for Epstein-Barr Virus (EBV) by an EBNA method
13. Evidence of infiltrate, cavitation, or consolidation on chest x-ray during pre-study screening.
14. Schizophrenia, bipolar disorder, or major depression that is unstable or uncontrolled on current medications.
15. Ongoing substance abuse; drug or alcohol.
16. Recent history of noncompliance.
17. Any medical condition that, in the opinion of the investigator, will interfere with the safe completion of the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2000-09; Primary Completion 2004-09 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Assess the incidence and severity of hypoglycemia in type 1 diabetic subjects receiving an islet allotransplant and immunotherapy during the first year posttransplant. | 1 year
Assess liver laboratory tests during the first year following intraportal islet allotransplantation. | 1 yr
Assess the incidence, type, and severity of islet transplant-related infectious complications during the first year posttransplant. | 1 year
Assess the proportion of recipients who develop alloantibodies directed at donor alloantigens during the first year posttransplant. | 1 year
Monitor the incidence, timing, and severity of adverse events as well as their relationship to the islet transplant procedure and additional protocol-regulated treatment products during the first year after islet transplantation. | 1 year

SECONDARY OUTCOMES:
Assess the proportion of type 1 diabetic subjects receiving delayed mycophenolate mofetil instead of tacrolimus who achieve insulin independence in the first year after transplantation of allogeneic islets. | 1 year
Assess the proportion of type 1 diabetic islet allograft recipients with full and partial alloislet function at one year post transplant. | 1 year
Assess the glycemic control, insulin secretory responses, and the glucose disposal rate during the first year posttransplant. | 1 year
Effect of donor age, pretransplant islet insulin secretory response, # of transplanted islet equivalents, # of transplanted beta cells, pretransplant insulin action, recipient BMI and immunosuppressive therapy on safety and efficacy. | 1 year
Assess, in a selected group of islet allotransplant recipients, the autoimmune and alloimmune responses to transplanted islets at intervals during the first year posttransplant. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard J. Hering, M.D., Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Result] Hering BJ, Kandaswamy R, Ansite JD, Eckman PM, Nakano M, Sawada T, Matsumoto I, Ihm SH, Zhang HJ, Parkey J, Hunter DW, Sutherland DE. Single-donor, marginal-dose islet transplantation in patients with type 1 diabetes. JAMA. 2005 Feb 16;293(7):830-5. doi: 10.1001/jama.293.7.830. PMID 15713772
- See also: Diabetes Institute for Immunology and Transplantation - U of M — http://www.diabetesinstitute.org